CLINICAL TRIAL: NCT00739583
Title: Visibility of Site Marking for Surgical Time Out With Two Different Skin Preparation Solutions
Acronym: site marking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Simon Mears, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NA_00011971
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-06

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Skin preparation; Skin marking; site marking; Site identification
MeSH Terms: interventions — Chromogranins; Iodophors; DuraPrep; Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Skin preparation for hip replacement with a Chlorhexidine based skin preparation solution, Chloraprep® (CHG 2% w/v and IPA 70% v/v; Enturia Inc., Leawood, KS, USA)
  Interventions: Drug: CHG 2% w/v and IPA 70% v/v
- 2 (Active Comparator): Skin preparation for hip replacement with an Iodine based skin preparation solution, Duraprep® (Iodophor 0.7% and IPA 74% w/w; 3M Healthcare, St. Paul, MN, USA.
  Interventions: Drug: Iodophor 0.7% and IPA 74% w/w

INTERVENTIONS:
Drug: CHG 2% w/v and IPA 70% v/v — Skin preparation of the surgical site per label of the product. The area for surgery will be prepared for 30 seconds
  Other Names: Chloraprep® (CHG 2% w/v and IPA 70% v/v; Enturia Inc., Leawood, KS, USA)
  Arms: 1
Drug: Iodophor 0.7% and IPA 74% w/w — Skin preparation of the surgical site per product labeling. The area will be painted with the solution.
  Other Names: Duraprep® (Iodophor 0.7% and IPA 74% w/w; 3M Healthcare, St. Paul, MN, USA)
  Arms: 2

SUMMARY:
Skin preparation solutions are used to clean the skin of the patient before surgery to decrease the rate of infection. This is particularly important for hip replacement to reduce the risk of prosthetic joint infection. The use of a mark on the skin for site identification has become the standard of care to decrease wrong site surgery. The Joint Commission has mandated site identification as part of the surgical "time-out". This procedure is also mandated by hospital policy.

Preliminary work on cadaveric skin shows that the type of skin preparation can erase the mark used for surgical site identification. Erasure of the mark presents the surgeon with difficulty in performing the site identification. Any error or lack of visualization of the site marking could lead to catastrophic wrong site surgery.

The investigators hypothesis is that chlorhexidine based skin preparation solutions erase site marking in comparison to iodine based skin preparation solutions. The investigators intend to prospectively study twenty patients undergoing total hip arthroplasty. Patients will be randomized to either a chlorhexidine based or an iodine based skin preparation solution. These solutions are both the current gold standard of clinical care. No differences have been shown in infection rates for total hip arthroplasty between these solutions. The site marking will be performed by the same surgeon in a standardized manner. The site marking will include the surgeon's three initials as per usual routine. Underneath the initials three random initials will be placed with a horizontal line drawn underneath. The preparation of the skin will be performed according to the manufacturer's specifications. Digital photographs will be taken of the skin marking after skin preparation. Photographs of the three random initials will be de-identified and placed in a "Powerpoint" presentation form. Ten orthopaedic surgeons will then read the site markings to identify the random initials and to tell whether the mark looks appropriate to perform a surgical timeout. The horizontal line will be digitally analyzed using Adobe Photoshop to quantitatively measure blackness of the mark.

DETAILED DESCRIPTION:
Abstract:

Skin preparation solutions are used to clean the skin of the patient before surgery to decrease the rate if infection. This is particularly important for hip replacement to reduce the risk of prosthetic joint infection. The use of a mark on the skin for site identification has become the standard of care to decrease wrong site surgery. The Joint Commission has mandated site identification as part of the surgical "time-out". This procedure is also mandated by hospital policy. Preliminary work on cadaveric skin shows that the type of skin preparation can erase the mark used for surgical site identification. Erasure of the mark presents the surgeon with difficulty in performing the site identification. Any error or lack of visualization of the site marking could lead to catastrophic wrong site surgery. Our hypothesis is that chlorhexidine based skin preparation solutions erase site marking in comparison to iodine based skin marking solutions. We intend to prospectively study twenty patients undergoing total hip arthroplasty to determine if the site marking is erased by chlorhexidine based skin preparation solutions when compared to iodine based skin preparation solutions. This information is critical to all surgeons who must balance the risk of wound infection versus wrong site surgery.

Study Procedures:

We intend to study twenty patients of one orthopaedic surgeon (SCM) undergoing total hip replacement in the supine position. Patients must be English speaking and of light skin color to standardize the contrast of the site marking. The study will be discussed with the patient in the clinic setting before the surgical date. Patients will be randomized into either using a chlorhexidine based skin preparation solution (Chloraprep® (chlorhexidine gluconate 2% w/v and isopropyl alcohol 70% v/v; Enturia Inc., Leawood, KS, USA)), or an iodine based skin preparation solution (Duraprep® (Iodophor 0.7% and isopropyl alcohol 74% w/w; 3M Healthcare, St. Paul, MN, USA)). Patients with allergies to either chlorhexidine or iodine will not be included in the study. These solutions are both the current gold standard of clinical care and are routinely used in the Johns Hopkins Bayview Medical Center. No differences have been shown in infection rates for total hip arthroplasty between these solutions.

The site marking will be performed by the surgeon in a standardized manner using the standard marker supplied at the hospital (Sharpie Fine Point Permanent Marker, Sanford Corporation, Oak Brook, IL, USA). All markings will be made in the pre-operative holding area per usual routine. The site marking will be made next to the site of the incision on the anterior thigh. The site marking will include the surgeon's three initials as per usual routine. Underneath the surgeon's initials, three random initials will be placed with a horizontal line drawn underneath. Twenty random three-letter combinations will be pre-generated using MS Excel® (Microsoft Office 2003, Microsoft Corporation, Seattle WA).

After patient positioning and prior to skin preparation an extra surgical time-out and site identification will be performed. The preparation of the skin will then be conducted according to the manufacturer's specifications for each skin preparation solution. After skin preparation, the solution will be allowed to dry while the patient is draped. Prior to applying the impermeable drape to the skin, digital photographs will be taken. Specimens will be photographed using a digital still camera (Digital Rebel XTi, Canon U.S.A., Lake Success, NY) with a 100-mm macro lens (EF 100mm f/2.8 USM Macro Lens, Canon U.S.A.), and ring flash (MR-14EX TTL, Canon U.S.A). The camera captures data at 10.1 megapixels and will be set in RAW mode. The shutter speed will be set at 1/60s with an F-stop value of 4.0. The camera was placed at a fixed distance from the skin using a tripod. After photography the impervious drape will be placed and another surgical time-out will be performed. The surgeon, anesthesiologist and nurse must all agree on the surgical site and it must be confirmed with the consent form, the patient records and the radiographs.

The study will make no changes in the clinic care of the patient besides the use of an additional time-out and the extra initials and the photograph of the site marking. The surgical procedure will not be altered in any way.

Photographs of the three random initials will be de-identified. They will be cropped using Adobe Photoshop CS2® (Adobe, San Jose, CA) so that only the three random initials and the horizontal line are visible. The file will be identified by a study number only. The files will be placed into a digital presentation (Powerpoint, Microsoft Office 2003, Microsoft Corporation, Seattle, WA). Ten orthopaedic surgeons will then read the site markings in random order. The surgeons will be asked to identify the initials and to tell whether the mark looks appropriate for them to perform a surgical timeout. The horizontal line will be digitally analyzed using Adobe Photoshop CS2® to quantitatively measure the mean gray level of the horizontal line using the histogram tool.

Regression analysis will be performed to examine the affect of the skin preparation solution on the ability of surgeons to correctly read the initials and their ability to identify the site marking.

Drugs/Substances/Devices:

Two skin preparation solutions will be used for this study. Both are considered gold standards for skin preparation and are routinely used at the Johns Hopkins Bayview Medical Center. These include:

Chlorhexidine based skin preparation solution

Chloraprep® (chlorhexidine gluconate 2% w/v and isopropyl alcohol 70% v/v; Enturia Inc., Leawood, KS, USA)

Iodine based skin preparation solution

Duraprep® (Iodophor 0.7% and isopropyl alcohol 74% w/w; 3M Healthcare, St. Paul, MN, USA)

Study Statistics:

Primary Variables:

Identification of the random initials by the reviewing orthopaedic surgeons

Judgment of reviewing orthopaedic surgeons that the site marking is identifiable for them to perform site identification

The mean gray level of the horizontal line

Risks:

Surgical site infection: The skin preparation of the skin will be conducting using the two standard skin preparation solutions at the Johns Hopkins Bayview Medical Center. The preparation will be performed according to manufacturer's directions for the skin preparation solutions. The risk of infection should not be changed by this study. This study is not meant to investigate the rates of infection using the two preparation solutions.

Wrong site surgery: The standard protocol for site identification will be performed for all patients. The surgeon's initials will be identified during the time-out procedure. The time out will be performed by the nurse in the operating room according to the protocol of the Johns Hopkins Bayview Medical Center. The nurse will read the consent form, confirm the site identification mark with the surgeon and the anesthesiologist. The side will be confirmed with the radiographs and the consent form for the procedure. The time out will be performed two times to prevent any possibility of wrong site surgery. This is a technique used by the neurosurgical services where site marking is difficult. The site will be identified both before and after the skin preparation.

Extra markings: The patient will have three extra initials and one horizontal line drawn underneath the standard site marking. Site markings are with permanent marker and do take several weeks of washing to be removed. All patients will be informed of the extra markings as part of the study consent form. If patients do not want to have these extra markings, they will not be included into the study.

Confidentiality:

The data from this study includes only the digital photographs of the site marking. The photographs will have no identifying information and will be only labeled with the study number (one to twenty). All information from this study will be de-identified data that should not pose any confidentiality risks to the patient.

Benefits:

The benefit of this study will be to give more information about the removal of site markings by skin preparation solutions. While the risk of wrong site surgery is currently low, everything possible must be done to eliminate any potential for this occurring. This study examines the marking used for total hip surgery; the risk of wrong site surgery is higher for those surgeries involving the digits or smaller areas of the body. In these areas, the marking must be perfect. Any elimination of the mark could result in catastrophe. If a mark is not well visible or partially erased, a culture is created where the mark is ignored, creating danger to the patient. If this is occurring with standard skin preparation solutions then either the solutions or the marking must be changed in the future. We hope that this study will help to eliminate any potential for wrong site surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Patients undergoing primary total hip surgery in a supine position.
* Patients must be of light skin color
* Patients must not be allergic to chlorhexidine or iodine

Exclusion Criteria:

* Non English speaking
* Patients not undergoing primary total hip surgery in a supine position.
* Patients not of light skin color
* Patients allergic to chlorhexidine or iodine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon c Mears, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Mears SC, Dinah AF, Knight TA, Frassica FJ, Belkoff SM. Visibility of surgical site marking after preoperative skin preparation. Eplasty. 2008 Jul 16;8:e35. PMID 18709136

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Group: Skin preparation for hip replacement with a Chlorhexidine based skin preparation solution, Chloraprep® (CHG 2% w/v and IPA 70% v/v; Enturia Inc., Leawood, KS, USA)
- Iodine Group: Skin preparation for hip replacement with an Iodine based skin preparation solution, Duraprep® (Iodophor 0.7% and IPA 74% w/w; 3M Healthcare, St. Paul, MN, USA.
Period: Overall Study
Arm/Group | Chlorhexidine Group | Iodine Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Group | Iodine Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (4.6) | 73 (4.2) | 72 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Identification of the Random Initials by the Reviewing Orthopaedic Surgeons
Description: The number of correctly identified initials as viewed by the orthopaedic surgeons. 10 participants were randomized to each study group. Each patient was marked with three initials. Each was viewed by ten surgeons giving a total of 300 initials for each group.
Time Frame: at time of surgery, approximately 10 minutes
Measure: Number; unit: number of correctly identified initals
Units Other Than Participants: number of random initials
Arm/Group | Chlorhexidine Group | Iodine Group
Number analyzed (Participants) | 10 | 10
Number analyzed (number of random initials) | 300 | 300
number of correctly identified initals | 209 | 296

2. Secondary Outcome: The Mean Change in Gray Level (Contrast) of the Horizontal Line
Description: The Mean change in gray level of the ink line as expressed in units between pre and post skin preparation. Gray level is a unitless value from 0-255 describing the brightness of a pixel (0 being black and 255 being white).
Time Frame: at time of surgery, approximately ten minutes
Measure: Mean (Standard Deviation); unit: gray level units
Units Other Than Participants: change in gray level
Arm/Group | Chlorhexidine Group | Iodine Group
Number analyzed (Participants) | 10 | 10
Number analyzed (change in gray level) | 10 | 10
gray level units | 59.8 (59.8) | 14.9 (11.4)

3. Secondary Outcome: Judgment of Reviewing Orthopaedic Surgeons That the Site Marking is Identifiable for Them to Perform Site Identification
Description: The number of sets of initials judged by the viewing orthopedic surgeons as sufficient for adequate site identification. Each participant was labeled with three initials to simulate a surgeon's initials. Ten orthopaedic surgeons determined if the initials were visible enough to allow for site identification. Each surgeon viewed all of the sets of initials, resulting in 100 viewed sets of initials in each group.
Time Frame: at time of surgery, approximately ten minutes
Measure: Number; unit: sets of intials
Units Other Than Participants: sets of initials
Arm/Group | Chlorhexidine Group | Iodine Group
Number analyzed (Participants) | 10 | 10
Number analyzed (sets of initials) | 100 | 100
sets of intials | 56 | 95

ADVERSE EVENTS:
Arm/Group | Chlorhexidine Group | Iodine Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Non-standardization of the amount of ink used to mark each site.

The use of only one type of marking pen.

No measurement of the amount of pressure use to apply the skin cleaning solutions.

Potential subjectivity of surgeons viewing initials

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No